CLINICAL TRIAL: NCT01375400
Title: Laboratory Effect on Platelet Activity of the First 300 mg Oral Dose Aspirin at the Acute Phase of Cerebral Ischemic Event.
Brief Title: Effect of Aspirin at the Acute Phase of Cerebral Ischemic Event.
Acronym: Aspirin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Direction recherche et innovation CHU Nancy, CentralHNF
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Aspirin
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Ischemic Stroke
Keywords: aspirin; platelet
MeSH Terms: conditions — Ischemic Stroke | interventions — Aspirin; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aspirin — Administration of 300 mg of aspirin, per os.
Biological: blood sample — 2 blood samples will be performed

SUMMARY:
Aspirin is the only anti-platelet medication used at the acute phase of ischemic stroke. The investigators would like to study laboratory effect of the first oral 300 mg dose of aspirin, given at hospital, after an ischemic event.

The principal hypothesis is that platelet activity would be able to recover during this day and could lead to ischemic recurrences.

Two blood samples are accomplished. The first 2 hours after aspirin intake and the second 23 hours after. Photometric aggregometry are performed with arachidonic acid and collagen induced platelet aggregation, measure of thromboxan B2 levels and reticular platelets count.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women
* Ischemic stroke less than 48 hours
* Signed consent

Exclusion Criteria:

* Danger to prescription of aspirin (haemorrhagic risk...)
* Prescription of heparin or VKA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Measure of platelet activity recovery within 24 hours after the first 300 mg oral dose of aspirin given at hospital at the acute phase of ischemic stroke | 1 month
  We study laboratory parameters of the first 300 mg oral dose of aspirin given, within 48 hours, after ischemic cerebral event. For all patients, two blood sampling are performed, the first, during the third hour after aspirin intake and the second during the twenty-fourth hour. Platelet reactivity is studied on the basis of serum thromboxane B2 levels and light transmission aggregometry after stimulation of platelet-rich plasma by acid arachidonic and collagen 2µg/ml reported to results with collagen 20 µg/ml.

SECONDARY OUTCOMES:
Measure of effect of the first 300 mg oral dose of aspirin given at the acute phase of cerebral ischemic stroke for already aspirin treated | 1 month
  For patients already treated with a daily dose of aspirin, a supplementary withdrawn was done before aspirin intake. Platelet reactivity was studied on the basis of serum thromboxane B2 levels and light transmission aggregometry after stimulation of platelet-rich plasma by acid arachidonic and collagen 2µg/ml reported to results with collagen 20 µg/ml.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital central, Nancy, France